CLINICAL TRIAL: NCT05540210
Title: Analytical Validation of the abioSCOPE Device With the IVD CAPSULE PSP Test: Comparison of PSP Values Measured With Venous Whole Blood and Those Measured With Arterial Whole Blood
Brief Title: Analytical Validation of the abioSCOPE Device With the in Vitro Device (IVD) CAPSULE PSP Test: Comparison of PSP Values Measured With Venous Whole Blood and Those Measured With Arterial Whole Blood
Acronym: AB-PSP-006
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI22_0021 (AB-PSP-006)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Stone Protein; Device
Keywords: Pancreatic Stone Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSP sample (Experimental)
  Interventions: Device: measurement of PSP

INTERVENTIONS:
Device: measurement of PSP — one or two blood samples

SUMMARY:
Abionic society has developed a novel point-of-care (POC) platform, the abioSCOPE, and an in vitro diagnostic kit for the quantification of the pancreatic stone protein (PSP) to be analyzed specifically with the abioSCOPE® device. The PSP is a host protein biomarker produced by the pancreas in response to a sepsis-related organ dysfunction and has shown a great potential in the early identification of septic patients This test is intended to be used to aid in the early recognition of sepsis. The test is extremely easy to use and has a total turnaround time of approximately 8 minutes. This test uses only 50 microliters of K2/K3-EDTA venous anticoagulated whole blood. Results are quantitative (ng/ml). The product is for Investigational Use Only in the US and bears CE-marking. It is commercially available in selected European and non-European countries. The test has also been clinically validated in a multicentric, prospective, observational study performed (AB-PSP-001, clinicaltrials.gov identifier NCT03474809).

The main goal of this study is to evaluate the analytical performances components of this product in a point-of-care environment, in particular the sample type comparability between arterial and venous whole blood.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated written informed consent by patient or close / family / trusted person prior to any mandatory study-specific procedures, sample collection, or analysis;
2. Male or female, 18 years of age or older;
3. Patient admitted to hospital
4. Need for venous and arterial blood samples as part of standard of care
5. Covered by a social security scheme.

Exclusion Criteria:

1. Subject suffering from a hematological pathology (coagulation disorder, severe anemia) that could interfere with the blood draw procedure;
2. Subject under juridical protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
PSP measurement | Day 1
  Pairwise comparability of test results when performed with K2-EDTA anticoagulated venous whole blood or K2-EDTA anticoagulated arterial whole blood, represented as percent recovery of arterial whole blood compared to venous whole blood, as well as scatter plots with Weighted Deming and Passing Bablok Regression, and bias plots.

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France